CLINICAL TRIAL: NCT01076660
Title: Left Ventricular Structural Predictors of Sudden Cardiac Death [Substudy of: Functional Energetics and Imaging for Phenotypic Characterization of Patients at Risk for Sudden Cardiac Death, See Also NCT000181233]
Brief Title: Left Ventricular Structural Predictors of Sudden Cardiac Death
Status: Recruiting | Type: Observational
Sponsor: Johns Hopkins University (Other)
Collaborators: Donald W. Reynolds Foundation (Other); Christiana Care Health Services (Other)
Responsible Party: Sponsor
Other Study IDs: IRB00324567
Record Dates: First submitted 2010-02-25; First posted 2010-02-26 (Estimated); Last update posted 2026-01-20 (Actual); Status verified 2026-01

CONDITIONS: Ischemic Cardiomyopathy; Nonischemic Cardiomyopathy
Keywords: Ischemic cardiomyopathy; Nonischemic cardiomyopathy; Implantable cardioverter defibrillator; Sudden Cardiac Death; Ventricular tachycardia; Ventricular fibrillation
MeSH Terms: conditions — Death, Sudden, Cardiac; Tachycardia, Ventricular; Ventricular Fibrillation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Sudden cardiac death (SCD) poses a significant health care challenge with high annual incidence and low survival rates. Implantable cardioverter defibrillators (ICDs) prevent SCD in patients with poor heart function. However, the critical survival benefit afforded by the devices is accompanied by short and long-term complications and a high economic burden. Moreover, in using current practice guidelines of reduced heart function, specifically left ventricular ejection fraction (LVEF)≤35%, as the main determining factor for patient selection, only a minority of patients actually benefit from ICD therapy (<25% in 5 years). There is an essential need for more robust diagnostic approaches to SCD risk stratification.

This project examines the hypothesis that structural abnormalities of the heart itself, above and beyond global LV dysfunction, are important predictors of SCD risk since they indicate the presence of the abnormal tissue substrate required for the abnormal electrical circuits and heart rhythms that actually lead to SCD. Information about the heart's structure will be obtained from cardiac magnetic resonance imaging and used in combination with a number of other clinical risk factors to see if certain characteristics can better predict patients at risk for SCD.

DETAILED DESCRIPTION:
Sudden cardiac death (SCD) poses a significant health care challenge with high annual incidence and low survival rates. Implantable cardioverter defibrillators (ICDs) prevent SCD in patients with left ventricular (LV) systolic dysfunction. However, the critical survival benefit afforded by the devices is accompanied by short and long-term complications and a high economic burden. Moreover, in using current practice guidelines of LV ejection fraction (LVEF)≤35% as the main determining factor for patient selection, only a minority of patients actually benefit from ICD therapy (<25% in 5 years). There is an essential need for more robust diagnostic approaches to SCD risk stratification.

This project examines the hypothesis that LV structural abnormalities above and beyond global LV dysfunction are important predictors of SCD risk since they indicate the presence of abnormal pathophysiologic substrate required for the ventricular arrhythmogenicity leading to SCD. This premise is supported by pre-clinical models and limited patient cohort studies examining the contribution of individual LV structural indices. However, there has been no prospective study of primary prevention ICD candidates in sufficiently large numbers to investigate the incremental value of a comprehensive assessment of LV structure on SCD risk over and above that of LVEF and readily available demographic and clinical variables.

LV structure can be quantified in detail using cardiac magnetic resonance imaging with late gadolinium enhancement (CMR-LGE). Specifically, accurate assessment of global LV function, volumes, mass, geometry, and infarct/scar characteristics are feasible and obtainable clinically in a single examination. We aim to examine whether or not any of these CMR indices or combination of indices are better able to discriminate between patients with high versus low susceptibility to SCD within the broader population of reduced LVEF patients. If the results of these studies demonstrate that LV structure is an important prognostic risk factor, it may be then be possible to more specifically focus ICD therapy to those who are most likely to benefit and avoid unnecessary device implantations.

ELIGIBILITY:
Inclusion Criteria:

* LVEF≤35%, referred clinically for ICD insertion for primary prevention purposes (i.e. no prior history of sustained ventricular arrhythmias)
* Between the ages of 21 and 80 years old
* Permission of the patient's clinical attending physician

Exclusion Criteria:

* Patients who refuse or are unable to give consent.
* Individuals with contraindications to MRI (i.e. implanted metallic objects such as pre-existing cardiac pacemakers, cerebral clips or indwelling metallic projectiles)
* Minors.
* Pregnant women.
* NYHA Class IV heart failure.
* Chronic renal insufficiency with creatinine clearance<60 ml/min; acute renal insufficiency of any severity
* Claustrophobia
* Prior adverse reaction to gadolinium-based contrast

Ages: 21 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with LV ejection fraction (LVEF) ≤35% of ischemic or nonischemic etiology (as measured by a clinical echocardiogram, ventriculogram, or radionuclide study) referred clinically for ICD insertion for primary prevention purposes (i.e. no prior history of sustained ventricular arrhythmias)
Sampling Method: Non-Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2003-10; Primary Completion 2028-06 (Estimated); Study Completion 2030-06 (Estimated)

PRIMARY OUTCOMES:
Composite SCD outcomes | Every 6 months for 5 years
  The first occurrence of an adjudicated appropriate ICD firing for ventricular tachycardia/ventricular fibrillation or cardiac death not treated by the ICD.

SECONDARY OUTCOMES:
Composite cardiac outcomes | Every 6 months for 5 years
  The first occurrence of an adjudicated appropriate ICD firing for ventricular tachycardia/ventricular fibrillation, hospitalization for heart failure or cardiac death.

CONTACTS AND LOCATIONS:
Overall Officials: Katherine Wu, MD, Principal Investigator — Johns Hopkins University
Locations (2):
- United States (2):
  - Christiana Care Health Services, Newark, Delaware
  - Johns Hopkins Medical Institutions, Baltimore, Maryland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Schmidt A, Azevedo CF, Cheng A, Gupta SN, Bluemke DA, Foo TK, Gerstenblith G, Weiss RG, Marban E, Tomaselli GF, Lima JA, Wu KC. Infarct tissue heterogeneity by magnetic resonance imaging identifies enhanced cardiac arrhythmia susceptibility in patients with left ventricular dysfunction. Circulation. 2007 Apr 17;115(15):2006-14. doi: 10.1161/CIRCULATIONAHA.106.653568. Epub 2007 Mar 26. PMID 17389270
- [Result] Fernandes VR, Wu KC, Rosen BD, Schmidt A, Lardo AC, Osman N, Halperin HR, Tomaselli G, Berger R, Bluemke DA, Marban E, Lima JA. Enhanced infarct border zone function and altered mechanical activation predict inducibility of monomorphic ventricular tachycardia in patients with ischemic cardiomyopathy. Radiology. 2007 Dec;245(3):712-9. doi: 10.1148/radiol.2452061615. Epub 2007 Oct 2. PMID 17911537
- [Result] Wu KC, Weiss RG, Thiemann DR, Kitagawa K, Schmidt A, Dalal D, Lai S, Bluemke DA, Gerstenblith G, Marban E, Tomaselli GF, Lima JA. Late gadolinium enhancement by cardiovascular magnetic resonance heralds an adverse prognosis in nonischemic cardiomyopathy. J Am Coll Cardiol. 2008 Jun 24;51(25):2414-21. doi: 10.1016/j.jacc.2008.03.018. PMID 18565399
- [Result] Ouwerkerk R, Bottomley PA, Solaiyappan M, Spooner AE, Tomaselli GF, Wu KC, Weiss RG. Tissue sodium concentration in myocardial infarction in humans: a quantitative 23Na MR imaging study. Radiology. 2008 Jul;248(1):88-96. doi: 10.1148/radiol.2481071027. PMID 18566171
- [Result] Ardekani S, Weiss RG, Lardo AC, George RT, Lima JA, Wu KC, Miller MI, Winslow RL, Younes L. Computational method for identifying and quantifying shape features of human left ventricular remodeling. Ann Biomed Eng. 2009 Jun;37(6):1043-54. doi: 10.1007/s10439-009-9677-2. Epub 2009 Mar 26. PMID 19322659
- [Result] Bottomley PA, Wu KC, Gerstenblith G, Schulman SP, Steinberg A, Weiss RG. Reduced myocardial creatine kinase flux in human myocardial infarction: an in vivo phosphorus magnetic resonance spectroscopy study. Circulation. 2009 Apr 14;119(14):1918-24. doi: 10.1161/CIRCULATIONAHA.108.823187. Epub 2009 Mar 30. PMID 19332463
- [Result] Strauss DG, Selvester RH, Lima JA, Arheden H, Miller JM, Gerstenblith G, Marban E, Weiss RG, Tomaselli GF, Wagner GS, Wu KC. ECG quantification of myocardial scar in cardiomyopathy patients with or without conduction defects: correlation with cardiac magnetic resonance and arrhythmogenesis. Circ Arrhythm Electrophysiol. 2008 Dec;1(5):327-36. doi: 10.1161/CIRCEP.108.798660. Epub 2008 Dec 2. PMID 19808427
- [Result] Strauss DG, Wu KC. Imaging myocardial scar and arrhythmic risk prediction--a role for the electrocardiogram? J Electrocardiol. 2009 Mar-Apr;42(2):138.e1-8. doi: 10.1016/j.jelectrocard.2008.12.010. Epub 2009 Jan 30. PMID 19185315
- [Result] Arevalo HJ, Vadakkumpadan F, Guallar E, Jebb A, Malamas P, Wu KC, Trayanova NA. Arrhythmia risk stratification of patients after myocardial infarction using personalized heart models. Nat Commun. 2016 May 10;7:11437. doi: 10.1038/ncomms11437. PMID 27164184
- [Result] Zhang Y, Guallar E, Weiss RG, Stillabower M, Gerstenblith G, Tomaselli GF, Wu KC. Associations between scar characteristics by cardiac magnetic resonance and changes in left ventricular ejection fraction in primary prevention defibrillator recipients. Heart Rhythm. 2016 Aug;13(8):1661-6. doi: 10.1016/j.hrthm.2016.04.013. Epub 2016 Apr 19. PMID 27108939
- [Result] Wu KC, Gerstenblith G, Guallar E, Marine JE, Dalal D, Cheng A, Marban E, Lima JA, Tomaselli GF, Weiss RG. Combined cardiac magnetic resonance imaging and C-reactive protein levels identify a cohort at low risk for defibrillator firings and death. Circ Cardiovasc Imaging. 2012 Mar;5(2):178-86. doi: 10.1161/CIRCIMAGING.111.968024. Epub 2012 Jan 20. PMID 22267750
- [Result] Sani MM, Sung E, Engels M, Daimee UA, Trayanova N, Wu KC, Chrispin J. Association of epicardial and intramyocardial fat with ventricular arrhythmias. Heart Rhythm. 2023 Dec;20(12):1699-1705. doi: 10.1016/j.hrthm.2023.08.033. Epub 2023 Aug 26. PMID 37640127
- [Result] Binder MS, Yanek LR, Yang W, Butcher B, Norgard S, Marine JE, Kolandaivelu A, Chrispin J, Fedarko NS, Calkins H, O'Rourke B, Wu KC, Tomaselli GF, Barth AS. Growth Differentiation Factor-15 Predicts Mortality and Heart Failure Exacerbation But Not Ventricular Arrhythmias in Patients With Cardiomyopathy. J Am Heart Assoc. 2023 Feb 7;12(3):e8023. doi: 10.1161/JAHA.122.026003. Epub 2023 Jan 31. PMID 36718879
- [Result] Vakil RM, Marine JE, Kolandaivelu A, Dickfeld T, Weiss RG, Tomaselli GF, Chrispin J, Wu KC. The Association of Clustered Ventricular Arrhythmia and Cycle Length With Scar Burden in Cardiomyopathy. JACC Clin Electrophysiol. 2022 Aug;8(8):957-966. doi: 10.1016/j.jacep.2022.05.008. Epub 2022 Jul 27. PMID 35981800
- [Result] Daimee UA, Sung E, Engels M, Halushka MK, Berger RD, Trayanova NA, Wu KC, Chrispin J. Association of left ventricular tissue heterogeneity and intramyocardial fat on computed tomography with ventricular arrhythmias in ischemic cardiomyopathy. Heart Rhythm O2. 2022 Apr 2;3(3):241-247. doi: 10.1016/j.hroo.2022.03.005. eCollection 2022 Jun. PMID 35734302
- [Result] Samuel TJ, Lai S, Schar M, Wu KC, Steinberg AM, Wei AC, Anderson ME, Tomaselli GF, Gerstenblith G, Bottomley PA, Weiss RG. Myocardial ATP depletion detected noninvasively predicts sudden cardiac death risk in patients with heart failure. JCI Insight. 2022 Jun 22;7(12):e157557. doi: 10.1172/jci.insight.157557. PMID 35579938
- [Result] Popescu DM, Shade JK, Lai C, Aronis KN, Ouyang D, Moorthy MV, Cook NR, Lee DC, Kadish A, Albert CM, Wu KC, Maggioni M, Trayanova NA. Arrhythmic sudden death survival prediction using deep learning analysis of scarring in the heart. Nat Cardiovasc Res. 2022 Apr;1(4):334-343. doi: 10.1038/s44161-022-00041-9. Epub 2022 Apr 7. PMID 35464150
- [Result] Popescu DM, Abramson HG, Yu R, Lai C, Shade JK, Wu KC, Maggioni M, Trayanova NA. Anatomically informed deep learning on contrast-enhanced cardiac magnetic resonance imaging for scar segmentation and clinical feature extraction. Cardiovasc Digit Health J. 2021 Nov 26;3(1):2-13. doi: 10.1016/j.cvdhj.2021.11.007. eCollection 2022 Feb. PMID 35265930
- [Result] Krebs J, Mansi T, Delingette H, Lou B, Lima JAC, Tao S, Ciuffo LA, Norgard S, Butcher B, Lee WH, Chamera E, Dickfeld TM, Stillabower M, Marine JE, Weiss RG, Tomaselli GF, Halperin H, Wu KC, Ashikaga H. CinE caRdiac magneTic resonAnce to predIct veNTricular arrhYthmia (CERTAINTY). Sci Rep. 2021 Nov 22;11(1):22683. doi: 10.1038/s41598-021-02111-7. PMID 34811411
- [Result] Wu KC, Wongvibulsin S, Tao S, Ashikaga H, Stillabower M, Dickfeld TM, Marine JE, Weiss RG, Tomaselli GF, Zeger SL. Baseline and Dynamic Risk Predictors of Appropriate Implantable Cardioverter Defibrillator Therapy. J Am Heart Assoc. 2020 Oct 20;9(20):e017002. doi: 10.1161/JAHA.120.017002. Epub 2020 Oct 7. PMID 33023350
- [Result] Okada DR, Miller J, Chrispin J, Prakosa A, Trayanova N, Jones S, Maggioni M, Wu KC. Substrate Spatial Complexity Analysis for the Prediction of Ventricular Arrhythmias in Patients With Ischemic Cardiomyopathy. Circ Arrhythm Electrophysiol. 2020 Apr;13(4):e007975. doi: 10.1161/CIRCEP.119.007975. Epub 2020 Mar 18. PMID 32188287
- [Result] Wongvibulsin S, Wu KC, Zeger SL. Improving Clinical Translation of Machine Learning Approaches Through Clinician-Tailored Visual Displays of Black Box Algorithms: Development and Validation. JMIR Med Inform. 2020 Jun 9;8(6):e15791. doi: 10.2196/15791. PMID 32515746
- [Result] Wu KC. Sudden Cardiac Death Substrate Imaged by Magnetic Resonance Imaging: From Investigational Tool to Clinical Applications. Circ Cardiovasc Imaging. 2017 Jul;10(7):e005461. doi: 10.1161/CIRCIMAGING.116.005461. PMID 28637807
- [Derived] Wongvibulsin S, Wu KC, Zeger SL. Clinical risk prediction with random forests for survival, longitudinal, and multivariate (RF-SLAM) data analysis. BMC Med Res Methodol. 2019 Dec 31;20(1):1. doi: 10.1186/s12874-019-0863-0. PMID 31888507